CLINICAL TRIAL: NCT01715519
Title: A Double-blind, Placebo-controlled Randomized Trial of Vilazodone in the Treatment of Posttraumatic Stress Disorder
Brief Title: Vilazodone for the Treatment of Posttraumatic Stress Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Southern California Institute for Research and Education (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Michael Hollifield, MD, Director of Program for Traumatic Stress, Southern California Institute for Research and Education
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VII-IT-05
Record Dates: First submitted 2012-10-18; First posted 2012-10-29 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: PTSD; Depression
Keywords: Vilazodone; PTSD; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Therapeutics; Vilazodone Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Viibryd) (Experimental): 10 mg/day 1 to 7; 20 mg/day 8 to 14; 40 mg/day week 3 to end week 12. Subjects will then be tapered off vilazodone as follows: 20 mg/day week 13, 10 mg/day, week 14 and no medication during week 15.
  Interventions: Drug: Treatment (Viibryd)
- Placebo (Placebo Comparator): will be compared to the treatment group (viibryd)
  Interventions: Drug: Treatment (Viibryd)

INTERVENTIONS:
Drug: Treatment (Viibryd)
  Other Names: Vilazodone

SUMMARY:
The purpose of this study is to determine whether vilazodone is effective in the treatmen of Posttraumatic Stress Disorder (PTSD)and co-morbid mild or more depression.

ELIGIBILITY:
Inclusion Criteria:

* Participants must satisfy DSM-IV diagnostic criteria for chronic PTSD
* Evidence of PTSD disease base upon one or more of the following:
* Mild or greater depression on the Beck Depression Inventory -II (BDI-II, score> 12).
* May have other symptom co-morbid with PTSD (e.g., anxiety or somatic pain)
* Ability to comprehend and satisfactorily comply with protocol required and signed written informed consent prior to entering study procedure
* May be in psychotherapy if initiated at least three months prior to the screening visit. Subject must not discontinue or otherwise alter therapy during the study.
* Subject may not have taken any psychopharmacological medications within 7 days prior to Baseline visit.
* Negative urine pregnancy test at screening visit and for the duration of the study for women of childbearing potential.

Exclusion Criteria:

* Patients with a concurrent DSM-IV Axis I diagnosis in any of the following categories:

  1. Delirium, Dementia, Amnestic and other Cognitive disorders
  2. Lifetime Schizophrenia and other Psychotic Disorders
  3. lifetime Bipolar I Disorder
  4. Bipolar-II Disorder with an episode of hypomania within the last year
  5. Alcohol or Substance Dependence or Abuse (excluding nicotine) in one month prior to the Screening Visit
  6. Any other concurrent Axis I Disorder (including Major Depressive Disorder) must be secondary to the primary diagnosis of PTSD.
* Decisional incapacity (dementia)
* Use of centrally acting medications that potentially have an effect on biological expression
* Chronic pain levels requiring use of any opiate medications
* Known exposure to chemicals of physical traumas that cause neuropsychiatric sequelae
* Past chronic PTSD
* History of 2 or more treatment failures on SSRIs given primarily for the treatment of PTSD, in adequate does at the Investigator's opinion, for at least 8 weeks
* History of intolerance or hypersensitivity to SSRI's
* History of seizures
* Significant risk of committing suicide, or are homicidal or violent and in the Investigator's opinion in significant imminent risk of hurting others
* Treated with depot-neuroleptic within 3 months or MAO inhibitors within 30 day prior to Baseline visit
* Received ECT within 3 months prior to Screening visit
* Pregnant or nursing, women of childbearing potential who are sexually active and do not use adequate contraception, or who are judged to be unreliable in their use of contraception
* Positive urine drug screen, unless proven to be prescribed for a short-term course of treatment. Drug screen must be repeated at least 7 days after the last dose of prescription medication containing narcotics
* A medical condition, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial
* Requiring concomitant treatment with any psychotropic drug (except zolpidem for sleep)
* Plans to initiate or terminate any form of psychotherapy or behavior therapy during the study
* Receiving disability payments (> 50 % service connections or total Social Security) or who are involved in litigation for PTSD or other psychiatric illnesses.
* Unable to speak, read, and understand English or are judged by the investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2012-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PTSD symptoms | four months
  PCL-C
PTSD Diagnosis | 4 months
  CAPS

SECONDARY OUTCOMES:
Depression | four months
  BDI-II
Sleep | 4 months
  PSQI
Anxiety | 4 months
  HSCL-25

OTHER OUTCOMES:
Biomarkers | four months
  serum

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Veterans Affairs Long Beach Healthcare System, Long Beach, California
  - Veterans Affairs Nebraska Western-Iowa Healthcare Systems, Omaha, Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramaswamy S, Driscoll D, Reist C, Smith LM, Albers LJ, Rose J, Nguyen L, Monga V, Doria R, Hollifield M. A Double-Blind, Placebo-Controlled Randomized Trial of Vilazodone in the Treatment of Posttraumatic Stress Disorder and Comorbid Depression. Prim Care Companion CNS Disord. 2017 Aug 24;19(4):17m02138. doi: 10.4088/PCC.17m02138. PMID 28858440